CLINICAL TRIAL: NCT02651597
Title: A Randomized, Controlled, Cross-over Study of the Effect of Oats on Post Prandial Glucose Response
Brief Title: A Study of the Effect of Oats on Post Prandial Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B2015:142
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Normoglycemic; Normal Body Weight
Keywords: Oatmeal; Beta glucan; Postprandial Glycemic Response; Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Viscous (Experimental): Low Viscous Beta Glucan Oatmeal
  Interventions: Other: Oatmeal
- Medium Viscous (Experimental): Medium Viscous Beta Glucan Oatmeal
  Interventions: Other: Oatmeal
- High Viscous (Experimental): High Viscous Beta Glucan Oatmeal
  Interventions: Other: Oatmeal

INTERVENTIONS:
Other: Oatmeal

SUMMARY:
The objectives are to assess the effects of high viscosity vs. medium and low viscosity oat β-glucan on post-prandial glycemic response in healthy adult participants.

DETAILED DESCRIPTION:
The trial will be a 3 week double-blinded, randomized, cross-over design with 3 treatment intervention (oatmeal breakfasts costain low, medium and high viscosity of beta glucan) periods separated by about 5-7 days washout period. Normoglycemic (<5.6 mmol/L) males and females (12 of each) of age 18-45 y with a body mass index (BMI) of 18.5-29.9 kg/m2 will be recruited.

Each participant will receive each of the following breakfast foods in a random order: 1) oat meal containing low viscosity beta glucan; 2) oat meal containing medium viscosity beta glucan; 3) oat meal containing high viscosity beta glucan. The participants will be asked to consume one of the breakfast foods during each visit.

Following each blood sample, appetite, physical comfort, energy/fatigue, and palatability of treatments will be measured by visual analogue scales (VAS).

Glucose measurements: Capillary blood will be collected during each visit by finger prick. Blood will be collected at fasting and at 15, 30, 45, 60, 90 and 120 minutes after the first bite/sip of the test product according to the Clinical Laboratory Standard Institute (CLSI) guidelines. Blood glucose will be measured in finger prick blood samples by glucose meters .

Males will be scheduled for three sessions over 3 weeks. Women will be scheduled during the first two weeks of their menstrual cycle (follicular phase), once per week.

During the wash-out days (5 - 7 days between each phase), participants can go about their daily activities unrestricted with the following exception: no strenuous activity or alcohol consumption on the days before the clinic visit. The investigators will ask that participants go to sleep at the same time on the days before the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L)
* BMI= 18.5-29.9 kg/m²

Exclusion Criteria:

* A change in medication (dose or type) or medical event requiring hospitalization within the past month.
* Daily tobacco use.
* Eat meals at irregular or unusual times.
* Food allergy, aversion or unwillingness to eat study foods.
* Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect blood sugar.
* Presence of a gastrointestinal disorder.
* Currently pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 0-200 mins
  Total area under the curve (iAUC, mmol*min/L) for glucose

SECONDARY OUTCOMES:
Appetite (visual analogue scales) | 0-200 mins
  Measured by VAS questionnaire at 12 time points used to calculate area under curve
Physical Comfort | 0-200 mins
  Measured by VAS questionnaire at 12 time points used to calculate area under curve
Energy/Fatigue | 0-200mins
  Measured by VAS questionnaire at 12 time points used to calculate area under curve
Palatability | at 5 mins
  Measured by VAS questionnaire at 12 time points used to calculate area under curve

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada